CLINICAL TRIAL: NCT02377856
Title: Peginterferon Plus Ribavirin Combination Therapy for Hepatitis C Six Months After Onset of Acute Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ming-Lung Yu, MD. PhD., Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-960056; KMUH (Other: KMUH)
Record Dates: First submitted 2014-09-09; First posted 2015-03-04 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Acute Hepatitis C
Keywords: acute hepatitis C; treatment; SVR
MeSH Terms: interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): 40 patients will receive pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 24 weeks combination treatment, followed by 24 weeks of follow-up. 'pegylated interferon alpha 2a, ribavirin'
  Interventions: Drug: pegylated interferon alpha 2a, ribavirin
- observation (No Intervention): 40 patients without treatment will be followed for the clinical course for 1.5 year

INTERVENTIONS:
Drug: pegylated interferon alpha 2a, ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 24 weeks, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: intervention

SUMMARY:
Patients with acute hepatitis C virus (HCV) infection usually become chronicity if viremia persists after 6 months of infection. The result of using pegylated interferon plus ribavirin combination therapy upon these patients remains to be explored

DETAILED DESCRIPTION:
Combination therapy with pegylated interferon-alpha plus ribavirin has greatly improved the treatment efficacy and is the mainstream of treatment for chronic hepatitis C infection. Current guideline suggests pegylated interferon monotherapy for patients with acute HCV infection. The efficacy might greatly improves if the treatment starts earlier. An estimation of 20 percents of patients could recover from acute infection spontaneously within 6 months after exposure,however. The present study aims to clarify the efficacy of pegylated interferon and ribavirin combination therapy for patients with hepatitis C six months after onset of acute infection

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18-80 years of age
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA for > 6 months
* Compensated liver disease
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Present therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Clinical evidence or history of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption>40 g/day) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hgb <11 g/dL in women or <12 g/dL in men at screening
* Any patient with major thalassemia
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* Local or Systemic malignancy unstable status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
treatment efficacy in terms of SVR rate | 1.5 yr
  Efficacy - Sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period.

SECONDARY OUTCOMES:
safety issues regarding adverse events | 1.5 yrs
  patient safety of pegylated interferon and ribavirin combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung, Taiwan., Kaohsiung City, Taiwan